CLINICAL TRIAL: NCT01723189
Title: Central Apnoeas in the Course of Transient Ischemic Attack/Ischemic Stroke: Clinical, Prognostic, Pathophysiological Elements.
Brief Title: Pathophysiology of Central Apnoeas in Stroke Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: MPons (Other Government)
Collaborators: Advisory Board of scientific Reserch Ente Ospedaliero Cantonale, ABREOC (Unknown); University of Geneva, Switzerland (Other); University of Milan (Other)
Responsible Party: Sponsor-Investigator, MPons, Professor, Ospedale Civico, Lugano
Organization: Ospedale Civico, Lugano (Other Government)
Other Study IDs: EOC.NSI.12.04
Record Dates: First submitted 2012-10-19; First posted 2012-11-07 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: Central Apnoeas; Stroke Patients
Keywords: central apnoeas; stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Central Apnoeas Patients: • 30 patients diagnosed with TIA / ischemic stroke within 7 days of admission and evidence at polysomnography of central apnoea (central apnoea index> 10 / h, or Cheyne-Stokes breathing for more than 30% of total sleep time or mixed apneas with central apnoeas> 50% of total apneas)
- Obstructive apnoea patients: • 30 patients diagnosed with TIA / ischemic stroke within 7 days of admission and evidence at polysomnography of obstructive sleep apnea (apnea-hypopnea index> 20 / h)
- No SDB patients: * • 30 patients diagnosed with TIA / stroke within 7 days of admission and no evidence of sleep respiratory disorders at polysomnography
- Healthy controls: • 30 healthy controls matched for age, sex, race and BMI.

SUMMARY:
40% of patients with Sleep Disorder Breathing (SDB) appearing during the acute phase of stroke show a respiratory pattern characterized by central apnoeas and/or periodic breathing.

Clinical studies conducted in patients with hearth failure and central apnoeas have demonstrated the pathogenetic central role of hypersensitivity of central and peripheral chemoreceptors in association with baroreflex hypersensitivity, expression of hyperactivity of sympathetic nervous system.

The joint study of chemoreflexes and baroreflexes in patients with central apneas during the acute and subacute phase of ischemic stroke represents, to our knowledge, a novelty in literature, that should supply useful elements to clarify the pathogenesis and the clinical and prognostic significance of these disorders.

Investigators expect a difference in the analysis of the baroreflexes and chemoreflexes in patients with ischemic stroke/transient ischemic attack (TIA) and central apnoeas than patients with ischemic stroke not accompanied by respiratory problems and compared with healthy controls.

DETAILED DESCRIPTION:
Investigators expected to include in the study of 120 patients, aged between 35 and 75 years, belonging to the following diagnostic categories:

* 30 patients diagnosed with TIA / ischemic stroke within 7 days of admission and evidence at polysomnography of central apnoea (central apnoea index> 10 / h, or Cheyne-Stokes breathing for more than 30% of total sleep time or mixed apneas with central apnoeas> 50% of total apneas)
* 30 patients diagnosed with TIA / ischemic stroke within 7 days of admission and evidence at polysomnography of obstructive sleep apnea (apnea-hypopnea index> 20 / h)
* 30 patients diagnosed with TIA / stroke within 7 days of admission and no evidence of sleep respiratory disorders at polysomnography
* 30 healthy controls matched for age, sex, race and BMI.

For the study of the baroreflexes, patients will be subjected to continuous monitoring of ECG, beat-to-beat blood pressure measured at the finger by Portapress system, respiratory rate and ventilation by pneumotachograph. The tests will be performed in the supine position and then repeated in a sitting position. Data from such monitoring will be used for analysis of the harmonic components of the cardiac rate (RR interval) and the variability of blood pressure and respiratory rate, through the method of auto regressive analysis.

For the study of central chemoreceptors, investigator will use the steady-state hypercapnic test, which measures the ventilatory response to hypercapnia at a constant level of Oxygen partial pressure (PaO2). The ventilatory response to hypercapnia is calculated by the method of linear regression and is represented by the angular coefficient of the straight line that describes the variation of ventilation for each variation of alveolar carbon dioxide partial pressure (PCO2).

For the study of peripheral chemoreceptors will be used the single-breath or transient hypercapnia test. The patient makes a single deep breath of a gas mixture containing 85% O2 and 15% CO2 and then resume normal breathing. It is expected, therefore, a period of 3 seconds, required because the gases contained in the mixture may come from the pulmonary circulation to the peripheral circulation, at the level of peripheral chemoreceptors. The ventilation is recorded within the next 20-30 seconds, because in this time interval is evaluated only the sensitivity of the peripheral chemoreceptors, being the latency of response of the central chemoreceptors greater than 1 minute.

ELIGIBILITY:
Inclusion Criteria:

* Patients

  * ≥35 years old and < 75 years old
  * with clinical diagnosis of TIA or ischemic stroke
  * admitted in a Stroke Unit within 2 days from onset of symptoms
  * signed Informed Consent

Exclusion Criteria:

* Patients

  * with unstable clinical situation (cardio-respiratory or life-threatening medical conditions)
  * currently on continuous positive airway pressure (CPAP) or on CPAP during the last 3 months before stroke
  * with non-ischemic events (intracerebral/subarachnoid haemorrhage)
  * Patients with coma/stupor

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Baroreflexes | 3 months
  For the study of the baroreflexes, patients will be subjected to continuous monitoring of ECG, beat-to-beat blood pressure measured at the finger by Portapress system, respiratory rate and ventilation by pneumotachograph. The tests will be performed in the supine position and then repeated in a sitting position. Data from such monitoring will be used for analysis of the harmonic components of the RR interval and the variability of blood pressure and respiratory rate, through the method of auto regressive analysis.
Chemoreflexes | 3 months
  For the study of central and peripheral chemoreceptors, investigator will use the steady-state hypercapnic test, which measures the ventilatory response to hypercapnia at a constant level of PaO2, and the single-breath test in wich the subject makes a single deep breath of a gas mixture containing 85% O2 and 15% CO2 and then resume normal breathing. The ventilation is recorded within the next 20-30 seconds, because in this time interval is evaluated only the sensitivity of the peripheral chemoreceptors, being the latency of response of the central chemoreceptors greater than 1 minute.

SECONDARY OUTCOMES:
Apnoea-hypopnoea index (AHI) | 3 months
  Assessing prognosis and spontaneous temporal evolution of central apnoeas in patients with cerebral ischemic events.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Pons, MD, Principal Investigator — Ospedale Regionale di Lugano - Civico
Locations (1):
- Ospedale Civico, Lugano, Canton Ticino, Switzerland

REFERENCES:
- [Background] Bassetti CL. Sleep and stroke. Semin Neurol. 2005 Mar;25(1):19-32. doi: 10.1055/s-2005-867073. PMID 15798934
- [Background] Giannoni A, Emdin M, Poletti R, Bramanti F, Prontera C, Piepoli M, Passino C. Clinical significance of chemosensitivity in chronic heart failure: influence on neurohormonal derangement, Cheyne-Stokes respiration and arrhythmias. Clin Sci (Lond). 2008 Apr;114(7):489-97. doi: 10.1042/CS20070292. PMID 17961123
- [Background] Nopmaneejumruslers C, Kaneko Y, Hajek V, Zivanovic V, Bradley TD. Cheyne-Stokes respiration in stroke: relationship to hypocapnia and occult cardiac dysfunction. Am J Respir Crit Care Med. 2005 May 1;171(9):1048-52. doi: 10.1164/rccm.200411-1591OC. Epub 2005 Jan 21. PMID 15665317
- [Background] Siccoli MM, Valko PO, Hermann DM, Bassetti CL. Central periodic breathing during sleep in 74 patients with acute ischemic stroke - neurogenic and cardiogenic factors. J Neurol. 2008 Nov;255(11):1687-92. doi: 10.1007/s00415-008-0981-9. Epub 2008 Nov 13. PMID 19009334
- [Background] Robinson TG, James M, Youde J, Panerai R, Potter J. Cardiac baroreceptor sensitivity is impaired after acute stroke. Stroke. 1997 Sep;28(9):1671-6. doi: 10.1161/01.str.28.9.1671. PMID 9303008
- [Background] Eames PJ, Blake MJ, Dawson SL, Panerai RB, Potter JF. Dynamic cerebral autoregulation and beat to beat blood pressure control are impaired in acute ischaemic stroke. J Neurol Neurosurg Psychiatry. 2002 Apr;72(4):467-72. doi: 10.1136/jnnp.72.4.467. PMID 11909905
- [Background] Sykora M, Diedler J, Turcani P, Hacke W, Steiner T. Baroreflex: a new therapeutic target in human stroke? Stroke. 2009 Dec;40(12):e678-82. doi: 10.1161/STROKEAHA.109.565838. Epub 2009 Oct 15. PMID 19834010
- [Background] Yumino D, Bradley TD. Central sleep apnea and Cheyne-Stokes respiration. Proc Am Thorac Soc. 2008 Feb 15;5(2):226-36. doi: 10.1513/pats.200708-129MG. PMID 18250216
- See also: Homepage of study center — http://www.eoc.ch